CLINICAL TRIAL: NCT03134586
Title: A Comparative Study of the Diagnostic Validity of Ultrasound, Magnetic Resonance Imaging and Capsule Endoscopy of Both the Small and Large Intestine in Suspected Crohn's Disease
Brief Title: Advanced Non-Invasive Diagnostics in Inflammatory Bowel Disease
Acronym: ANDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Sygehus Lillebaelt (Other)
Responsible Party: Principal Investigator, Jacob Brodersen, Specialist Registrat, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ANDI 1
Record Dates: First submitted 2017-01-06; First posted 2017-05-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Crohn Disease
Keywords: Capsule endoscopy; Crohn's disease; Magnetic resonance enterography; Ileocolonoscopy; Bowel Ultrasound; diagnostic imaging
MeSH Terms: conditions — Crohn Disease | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- trial participant (Other): All participants undergoes the same diagnostic imaging
  Interventions: Other: Diagnostic imaging

INTERVENTIONS:
Other: Diagnostic imaging

SUMMARY:
The purpose of this study is to determine whether Non-invasive endoscopic procedures (pillcam colon capsule endoscopy, PCCE) and non-ionizing radiological modalities (MR enterocolonography, MREC and ultrasound, US) - offer a sufficiently high diagnostic validity in patients with suspected CD compared to the traditional invasive approach using ileocolonoscopy with biopsies as first line diagnostic modality

DETAILED DESCRIPTION:
This is a prospective, blinded, multicenter study of the diagnostic validity, inter-observer agreement, image quality and subjective experience of discomfort with PCCE, MREC and US in patients with suspected CD. Ileocolonoscopy serves as the diagnostic gold standard. Patients are recruited from 3 centers in the Region of Southern Denmark managing adult patients with inflammatory bowel diseases. Each patient goes through a standardized work-up including medical history, physical examination, C-reactive protein, fecal calprotectin, ileocolonoscopy, PCCE, MREC and US. All examinations are reviewed and described in a standardized fashion. The radiologists and physicians describing PCCE, MREC, and US are blinded to the findings at ileocolonoscopy and the other imaging modalities.

ELIGIBILITY:
Inclusion Criteria:

General criterion

All of the following:

* Clinical suspicion of CD
* Age > 15 years
* Negative serologic markers for celiac disease, negative stool culture (or polymerase chain reaction) for pathogenic bacteria and a negative microscopy for intestinal parasites
* Fecal calprotectin > 50 mg/kg
* Signed informed consent

Clinical criterion Diarrhea and/or abdominal pain for more than 1 month (or repeated episodes of diarrhea and/or abdominal pain) associated with one or more of the following findings: (1) C-reactive protein (CRP) >5 mg/L, (2) thrombocytosis (> 400 x 109/L), anemia (hemoglobin < 7.0 mmol/L for women and < 8.0 mmol /L for men or a decrease > 0.5 mmol/L compared to the usual level), (3) prolonged fever (> 37.5 C for more than 2 weeks), (5) weight loss (≥ 3 kg or ≥ 5% compared to the normal body weight), (6) perianal abscess/fistula, or (7) a family history of inflammatory bowel disease.

Exclusion Criteria:

* Acute bowel obstruction
* Intake of NSAIDs or acetylsalicylic acid ≤ 4 weeks before inclusion except prophylactic treatment with low dose Aspirin (≤ 150 mg per day)
* Pregnancy or lactation
* Alcohol or drug abuse
* Known gastrointestinal disorder other than inflammatory bowel disease
* Renal failure defined by a plasma-creatinine above the normal reference range
* Claustrophobia, cardiac pacemaker or implanted magnetic foreign bodies that precludes MREC
* Interpreter required or inability to understand the oral and written information
* Colonoscopy contraindicated, performed within 3 months or unwillingness to go through colonoscopy

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of PCCE, MREC and US for the diagnosis of CD | 36 months
  Sensitivity and specificity of PCCE, MREC and US for the diagnosis of CD located in the terminal ileum and colon (per patient & per segment). Ileocolonoscopy serves as gold standard
Correlation of disease severity | 36 months
  Correlation of disease severity assessed with PCCE, MREC, US and ileocolonoscopy
Inter-observer agreement | 36 months
  Inter-observer agreement with PCCE, MREC, US and ileocolonoscopy

SECONDARY OUTCOMES:
Diagnostic yield of proximal CD | 36 months
  Diagnostic yield of PCCE, MREC and US for CD located proximal to the terminal ileum
Patients reported experience | 36 months
  Patients' subjective experience of discomfort during PCCE, MREC, US and ileocolonoscopy
Interobserver PCCE | 36 months
  Sensitivity and specificity of PCCE with different reading protocols
Utility of diffusion weighed magnetic resonance imaging (dw-MREC) and US Doppler flow | 36 months
  Utility of diffusion weighed magnetic resonance imaging (dw-MREC) and US Doppler flow (Limberg score): Sensitivity, specificity and correlation with endoscopic disease activity

CONTACTS AND LOCATIONS:
Overall Officials: Jacob B Brodersen, MD, Principal Investigator — Esbjerg Hospital - University Hospital of Southern Denmark
Locations (3):
- Denmark (3):
  - Sydvestjysk sygehus, Esbjerg
  - Odense university Hospital, Odense
  - Sygehus Lillebaelt, Vejle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brodersen JB, Jensen MD, Juel MA, Kjeldsen J, Knudsen T, Rafaelsen SR. Intestinal ultrasound in patients with suspected Crohn's disease - results of a prospective evaluation by trainees. Scand J Gastroenterol. 2023 Jul-Dec;58(12):1405-1411. doi: 10.1080/00365521.2023.2234538. Epub 2023 Jul 17. PMID 37459054
- [Derived] Brodersen JB, Knudsen T, Kjeldsen J, Juel MA, Rafaelsen SR, Jensen MD. Diagnostic accuracy of pan-enteric capsule endoscopy and magnetic resonance enterocolonography in suspected Crohn's disease. United European Gastroenterol J. 2022 Nov;10(9):973-982. doi: 10.1002/ueg2.12307. Epub 2022 Sep 7. PMID 36069336